CLINICAL TRIAL: NCT04628598
Title: Effects of The Pregnant Follow-Up Conducted With Home Visits on The Perinatal Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayça Demir Yıldırım, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulUCAycaDemirYıldırım
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy Related; Prenatal Care Late
Keywords: Pregnancy; Home Visit; Antenatal Care; Perinatal Period; Antenatal; İnnatal; Postnatal
MeSH Terms: interventions — Prenatal Care; Prenatal Education

STUDY DESIGN:
Intervention Model Description: The experiment and control group will be put into study at the same time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home visiting pregnant women (Experimental): The pregnant women in the experimental group will be given education and care with home visits.
  Interventions: Behavioral: Antenatal care and prenatal education with a home visit
- Control Group (No Intervention): Home visits will not be made to the control group, only the primary care antenatal care will be followed.

INTERVENTIONS:
Behavioral: Antenatal care and prenatal education with a home visit — Providing prenatal education and care by home visits to pregnant women
  Arms: Home visiting pregnant women

SUMMARY:
The World Health Organization (WHO) developed a safe motherhood program in 1987 to reduce maternal and infant mortality. Safe motherhood is maximizing maternal and child health. This is only possible with the highest level of prenatal, delivery and postnatal care. Care has a priority and special place in primary health care services. It increases access to preventive services such as monitoring prenatal and postnatal follow-ups in primary care, pregnant, postpartum and newborn health, immunization, training and counseling, early detection of risk, and decreases unwanted consequences. Home visits are a non-pharmacological and priority method in prenatal care. With this method, when healthcare providers (nurses, midwives) provide healthcare services to women in their own homes, it ensures the support and development of prenatal, maternal, infant and child health together with social, psychological, economic, familial and other factors. Prenatal care in Turkey is such that there will be at least four follow-ups. Current antenatal care guides suggest more contact with pregnant women.

This study will examine the effects of pregnancy follow-up with home visits on perinatal outcomes.

DETAILED DESCRIPTION:
Implementing a home visit program during pregnancy is a comprehensive and important strategic step to prevent adverse birth outcomes during pregnancy. Studies in the literature suggest that care provided at home or by one-on-one healthcare personnel can encourage healthy prenatal behaviors with psychosocial support, social service and nutritional support. Home visit programs instead of standard antenatal care (ANC) have the potential to make a difference. For home visits to be effective, home visitors should not only inform women about the risks and values of certain behaviors, but also help them develop individualized strategies for behavior change.

The importance of home visits in prenatal pregnancy follow-up in the nineteen century has been demonstrated by many studies. Today, home visits are supported by studies in the literature, as it is a healthy start to life and a more promising model for reaching pregnant women. A Cochrane study published moderate evidence that women prefer flexible home visits rather than a rigid appointment system.

Turkey Demographic and Health Survey (DHS) prior to birth by the 2018 four and older care-taking rate in care increased by a certain momentum until 2013, there has been a significant change in the ratio between said from 2013 to 2018. Although the total fertility rate in Turkey is 2.3, it varies according to the regions. The age at marriage for adolescents is 15%, and the rate of becoming an adolescent mother is 4%. Delivery methods of women result in 54% of cesarean delivery. 29% of women are overweight and 30% are obese. Turkey Statistical Institute (TSI), according to the women's smoking rate was 13.1%. There are a limited number of studies reflecting the smoking status of pregnant women in the country. In a study conducted on this subject, the rate of smoking during pregnancy was reported as 37% of women who smoke before pregnancy. Considering the data on women's health and reproductive health, new models are needed for the provision of preventive health services that will realize the goals of "maternal mortality" and "healthy and quality life", which are among the sustainable development indicators of the country. Antenatal care is an important key for lowering the maternal mortality rate and for a healthy and quality life in pregnancy. Prenatal care in Turkey is such that there will be at least four follow-ups. Current antenatal care guidelines recommend more contact with pregnant women. Models are needed to monitor and increase the results of antenatal care. For Turkey, there is a need to present the 'Antenatal Care Guide' published by the Ministry of Health with a model designed in accordance with the data and culture of the country for primary care follow-up. There is currently no strong evidence that home visits improve the use of routine antenatal services, but most studies do not yet shed detailed light on this issue.

There are 50 different home visit models serving in different areas around the world. Main goals; to play a common role in maternal, child health and healthy shaping of parents' lives. Most of these models work on the basis of evidence. There are 16 models with maternal results. While some of the models have a very good effect on maternal outcome, there is research showing that some are lower. Each model also differs in terms of follow-up time and service providers. Some home visit patterns start with pregnancy and continue until the newborn is two years old, while some home visits may be shorter. Some models are run by nurses, some are assistant professionals in nurse supervision (a job title given to people who are trained but not professionally licensed to assist professionals in various professions such as education, health, engineering, and law) and non-professionals (mentor mothers who give birth and breastfeed) done by. In other models, social workers, psychologists, child mental health assistant specialists and / or assistant assistants in this field are managers.

In Turkey, ANC is among the routine services in order to increase the level of maternal health and reduce maternal mortality, and it is applied throughout the country. According to the "Antenatal Care Management Guideline", pregnant women are followed up at least four times if there is no risk. The guide recommends that each pregnant should be followed up for at least four times. It is recommended to perform once between 24 weeks, third follow-up between 28-32 weeks and fourth follow-up between 36-38 weeks.

Today's understanding of health in Turkey and developing countries still focuses on the treatment of diseases and patient care. However, nurses working in primary health care, preventive health care, healthy individuals and healthy families have taken important steps to develop individual family functionality. The duration, frequency and intensity of home visits raise many evidence-based results. It is among the results that it decreases the risks especially related to lifestyle and preterm birth. Home visits during the prenatal period are seen as a part of continuous and comprehensive health care that enables pregnant women and their families to be evaluated as a whole within their own living space. In Turkey, home visits to pregnant women were first started to be carried out by health centers with the socialization law of health in 1960, and especially the pregnant women were identified by home visits. The family medicine system was switched to the whole country in 2010 and a new system was introduced with the health transformation law. Home visits are defined in the Family Medicine Regulation, but there are deficiencies in practice.

In this context, the antenatal care process carried out in primary care is supported by pregnant home visits as a new model, increasing the satisfaction of women from the service procurement, getting qualified prenatal care and consequently reducing the risks, being educated about pregnancy and birth, postpartum periods, and normal birth. It will help the mother to be prepared, reduce depression and increase her self-efficacy in breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* The pregnant woman is primiparas.
* Detection of the pregnant woman in family medicine software
* The pregnant woman does not have a high risk pregnancy.
* Finding a single fetus in the pregnant woman.
* Not having received infertility treatment.
* The pregnant woman did not have a psychiatric diagnosis.
* The pregnant woman's acceptance to participate in the research.

Exclusion Criteria:

* Being in the high risk category of the pregnant woman
* The mother tongue is not Turkish
* Having attended a planned, periodic pregnancy school course
* Being multiparous

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Prenatal education knowledge rate | Thirteen(13) weeks
  During home visits, pregnant women will be given birth preparation training, and after the last training, pre-test-post-test questionnaires will be conducted regarding pregnancy, delivery and the postpartum period, and accurate information rates will be checked. In the questionnaire, the correct information status will be answered as correct, incorrect and I have no idea, and as the number of correct increases between the pre-test and post-test, the level of knowledge will be considered as higher.
Spontaneous vaginal birth rate | Eight (8) months
  After the home visits of pregnant women, a questionnaire will be applied in the postpartum period and delivery methods will be asked.
Breastfeeding Self-efficacy | Thirteen(13) weeks
  Breastfeeding Self-Efficacy Scale will be applied to look at the effect of breastfeeding training in the postpartum period during home visits during pregnancy.
  Breastfeeding Self-Efficacy Scale; Breastfeeding Self-Efficacy Scale is a 33-item scale developed by Dennis in 1999. It was first applied to 130 English-speaking Canadian women, the Cronbach alpha value was found to be 0.96, and the item-total correlation of 73% of the items was 0.30-0.70. He then developed the Brief Breastfeeding Self-Efficacy Scale by reducing the scale to a 14-item scale in 2003. Cronbach alpha value was found to be 0.94.
  Breastfeeding Self-Efficacy Short Form Scale is a 5-point Likert Type scale 1 = "Not sure at all" and 5 = "I'm always sure". As suggested by Bandura (1998), all items are in positive direction. The minimum score that can be obtained from the scale is 14 maximum 70. High score is an indicator of high breastfeeding self-efficacy.
Postpartum Depression | Thirteen(13) weeks
  Edinburgh Postpartum Depression Scale will be applied to examine the effect of home visits and prenatal education on postpartum depression.
  Edinburgh Postpartum Depression Scale (EPDS); EPDS is a 4-point Likert style self-report scale consisting of 10 items. PRES was adapted to Turkish by Engindeniz. In Engindeniz's validity and reliability study, this scale had an internal consistency coefficient of 0.79, a split-half reliability, a cut-off of 0.80 of 12/13, a sensitivity of 0.84, a specificity of 0.88, a positive predictive value of 0.69, and a negative predictive value of 0.94.
  The Edinburgh Postnatal Depression Scale is a 10-item self-report scale assessing the common symptoms of depression. Each item is scored on a 4 point scale (O-3), the minimum and maximum total score ranging from O-30, respec- tively.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Demir Yıldırım, Phd Student, Principal Investigator — Student
Locations (1):
- İstanbul Üniversitesi Cerrahpaşa, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not discussed and resolved among investigators

REFERENCES:
- [Background] Liu N, Li P, Wang J, Chen D, Sun W, Zhang W. Effects of home visits for pregnant and postpartum women on premature birth, low birth weight and rapid repeat birth: a meta-analysis and systematic review of randomized controlled trials. Fam Pract. 2019 Oct 8;36(5):533-543. doi: 10.1093/fampra/cmz009. PMID 30925194
- [Background] McLaughlin FJ, Altemeier WA, Christensen MJ, Sherrod KB, Dietrich MS, Stern DT. Randomized trial of comprehensive prenatal care for low-income women: effect on infant birth weight. Pediatrics. 1992 Jan;89(1):128-32. PMID 1727996
- [Background] Lee E, Mitchell-Herzfeld SD, Lowenfels AA, Greene R, Dorabawila V, DuMont KA. Reducing low birth weight through home visitation: a randomized controlled trial. Am J Prev Med. 2009 Feb;36(2):154-60. doi: 10.1016/j.amepre.2008.09.029. PMID 19135906
- [Background] Ichikawa K, Fujiwara T, Nakayama T. Effectiveness of Home Visits in Pregnancy as a Public Health Measure to Improve Birth Outcomes. PLoS One. 2015 Sep 8;10(9):e0137307. doi: 10.1371/journal.pone.0137307. eCollection 2015. PMID 26348847
- [Background] Downe S, Finlayson K, Tuncalp O, Gulmezoglu AM. Provision and uptake of routine antenatal services: a qualitative evidence synthesis. Cochrane Database Syst Rev. 2019 Jun 12;6(6):CD012392. doi: 10.1002/14651858.CD012392.pub2. PMID 31194903
- [Background] Stamuli E, Richardson G, Duffy S, Robling M, Hood K. Systematic review of the economic evidence on home visitation programmes for vulnerable pregnant women. Br Med Bull. 2015 Sep;115(1):19-44. doi: 10.1093/bmb/ldv032. Epub 2015 Jul 28. PMID 26224694
- [Background] Cluxton-Keller F, Donnelly CL, Williams M, Buteau J, Stolte P, Monroe-Cassel M, Bruce ML. An implementation-effectiveness hybrid trial of video-based family therapy for peripartum depression in home visited mothers: a protocol for a pilot trial. Pilot Feasibility Stud. 2017 Nov 13;3:55. doi: 10.1186/s40814-017-0203-2. eCollection 2017. PMID 29158913
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Background] Goyal NK, Hall ES, Meinzen-Derr JK, Kahn RS, Short JA, Van Ginkel JB, Ammerman RT. Dosage effect of prenatal home visiting on pregnancy outcomes in at-risk, first-time mothers. Pediatrics. 2013 Nov;132 Suppl 2(Suppl 2):S118-25. doi: 10.1542/peds.2013-1021J. PMID 24187113
- [Background] Alus Tokat M, Okumus H, Dennis CL. Translation and psychometric assessment of the Breast-feeding Self-Efficacy Scale-Short Form among pregnant and postnatal women in Turkey. Midwifery. 2010 Feb;26(1):101-8. doi: 10.1016/j.midw.2008.04.002. Epub 2008 Jun 9. PMID 18541350
- [Background] Korukcu O, Kukulu K, Firat MZ. The reliability and validity of the Turkish version of the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) with pregnant women. J Psychiatr Ment Health Nurs. 2012 Apr;19(3):193-202. doi: 10.1111/j.1365-2850.2011.01694.x. Epub 2012 Jan 20. PMID 22260727
- [Derived] Demir Yildirim A, Hotun Sahin N. Does Antenatal Care Integrate with Home Visits Effect Perinatal Outcomes? A Randomized Control Trial. Matern Child Health J. 2025 Dec 17. doi: 10.1007/s10995-025-04202-7. Online ahead of print. PMID 41407980
- See also: Review of Research on Home Visiting for Pregnant Women and Parents of Young Children. — https://www.researchgate.net/publication/237351287_Review_of_Research_on_Home_Visiting_for_Pregnant_Women_and_Parents_of_Young_Children
- See also: Universal progressive model oh home-visiting for pregnant women and young children at the primary health care level: Methodical recommendations for implementation in primary health care organizations — https://www.unicef.org/kazakhstan/sites/unicef.org.kazakhstan/files/2018-11/%D0%BC%D0%B5%D1%82%D0%BE%D0%B4%D0%B8%D1%87%D0%BA%D0%B0%20%D0%BD%D0%B0%20%D0%B0%D0%BD%D0%B3%D0%BB_FINAL_0.pdf
- See also: , 224 Sayılı Sağlık Hizmetlerinin Sosyalleştirilmesi Hakkında Kanun — https://www.mevzuat.gov.tr/MevzuatMetin/1.4.224.pdf
- See also: The Mother and Infant Home Visiting Program Evaluation-Strong Start: First Annual Report — https://www.mdrc.org/publication/first-annual-report-mother-and-infant-home-visiting-program-evaluation-strong-start
- See also: Guidelines for Perinatal Care. — https://www.acog.org/clinical-information/physician-faqs/-/media/3a22e153b67446a6b31fb051e469187c.ashx
- See also: Antenatal care for uncomplicated pregnancies, Clinical Guideline — https://www.nice.org.uk/guidance/cg62/resources/antenatal-care-for-uncomplicated-pregnancies-pdf-975564597445
- See also: Doğum Öncesi Ev Ziyareti Hizmeti Verilen Gebelerin Memnuniyet Düzeyleri — https://dergipark.org.tr/tr/pub/gumussagbil/issue/23826/253829